CLINICAL TRIAL: NCT07079631
Title: A Phase I/II, Randomized, Multi-site Trial to Investigate the Efficacy and Safety of BNT314 in Combination With BNT327 and Chemotherapy in Participants With Metastatic Colorectal Cancer
Brief Title: A Clinical Study to Test if an Investigational Treatment Called BNT314 When Used in Combination With Another Investigational Treatment BNT327 and Chemotherapy, is Beneficial and Safe for Patients With Advanced Colorectal Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Collaborators: Genmab (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BNT314-02; 2025-521768-36-00 (EU CTIS Number)
Record Dates: First submitted 2025-07-09; First posted 2025-07-23 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Microsatellite stable or mismatch repair proficient (MSS/pMMR) tumors; Immune checkpoint inhibitor; Programmed death-ligand 1 (PD-L1); Vascular endothelial growth factor-A (VEGF-A); Bispecific antibody; Immunotherapy; Combination chemotherapy; Dose optimization
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Masking Description: Part A and Part B of this study are open label. Only in Part C, the majority of sponsor personnel will be blinded to study treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Phase 1 (Part A): BNT314 (escalating dose levels) + BNT327 (Experimental): Up to 5 dose levels of BNT314. One or two dose levels of BNT327.
  Interventions: Biological: BNT314; Drug: BNT327
- Phase 1 (Part B): BNT314 + BNT327 + SoC chemotherapy 1 (Experimental): BNT314 (optimized dose level 1 or 2 as determined based on data from Part A) + BNT327 + SoC combination chemotherapy 1.
  One selected dose level of BNT327.
  Interventions: Biological: BNT314; Drug: BNT327; Drug: SoC chemotherapy treatment 1
- Phase 1 (Part B): BNT314 + BNT327 + SoC chemotherapy 2 (Experimental): BNT314 (optimized dose level 1 or 2 as determined based on data from Part A) + BNT327 + SoC combination chemotherapy 2.
  One selected dose level of BNT327.
  Interventions: Biological: BNT314; Drug: BNT327; Drug: SoC chemotherapy treatment 2
- Phase 2 (Part C): BNT314 + BNT327 + SoC chemotherapy 1 (Experimental): Recommended phase 2 dose of BNT314 + BNT327 + SoC combination chemotherapy 1. One selected dose level of BNT327.
  Interventions: Biological: BNT314; Drug: BNT327; Drug: SoC chemotherapy treatment 1
- Phase 2 (Part C): Bevacizumab + SoC chemotherapy 1 (Active Comparator): Combination of two different SoC therapies
  Interventions: Drug: SoC chemotherapy treatment 1; Drug: Bevacizumab
- Phase 2 (Part C): BNT327 + SoC chemotherapy 1 (Experimental): BNT327 + SoC combination chemotherapy 1. One selected dose level of BNT327.
  Interventions: Drug: BNT327; Drug: SoC chemotherapy treatment 1

INTERVENTIONS:
Biological: BNT314 — Intravenous (IV) infusion
  Arms: Phase 1 (Part A): BNT314 (escalating dose levels) + BNT327; Phase 1 (Part B): BNT314 + BNT327 + SoC chemotherapy 1; Phase 1 (Part B): BNT314 + BNT327 + SoC chemotherapy 2; Phase 2 (Part C): BNT314 + BNT327 + SoC chemotherapy 1
Drug: BNT327 — IV infusion
  Arms: Phase 1 (Part A): BNT314 (escalating dose levels) + BNT327; Phase 1 (Part B): BNT314 + BNT327 + SoC chemotherapy 1; Phase 1 (Part B): BNT314 + BNT327 + SoC chemotherapy 2; Phase 2 (Part C): BNT314 + BNT327 + SoC chemotherapy 1; Phase 2 (Part C): BNT327 + SoC chemotherapy 1
Drug: SoC chemotherapy treatment 1 — IV infusion / IV bolus
  Arms: Phase 1 (Part B): BNT314 + BNT327 + SoC chemotherapy 1; Phase 2 (Part C): BNT314 + BNT327 + SoC chemotherapy 1; Phase 2 (Part C): BNT327 + SoC chemotherapy 1; Phase 2 (Part C): Bevacizumab + SoC chemotherapy 1
Drug: SoC chemotherapy treatment 2 — IV infusion / IV bolus / oral
  Arms: Phase 1 (Part B): BNT314 + BNT327 + SoC chemotherapy 2
Drug: Bevacizumab — IV infusion
  Arms: Phase 2 (Part C): Bevacizumab + SoC chemotherapy 1

SUMMARY:
This randomized, multi-site, three-part study will test a new treatment called BNT314, which is designed to help the body's immune system fight cancer in combination with another new treatment (BNT327, which is an immune checkpoint inhibitor) and chemotherapy in participants with metastatic colorectal cancer (mCRC).

This study will enroll participants with microsatellite stable or mismatch repair proficient (MSS/pMMR) mCRC who did not respond well to their first schema of chemotherapy. In one part of the study (i.e., Part B) mCRC participants will be enrolled, who have not received any systemic therapy before for their cancer.

DETAILED DESCRIPTION:
The main study goals are as follows:

* Part A (Phase 1, safety run-in, dose escalation): To see if BNT314 in combination with BNT327 is safe for participants and to investigate if the administration of treatment that can be given safely, without causing severe side effects in participants.
* Part B (Phase 1, dose optimization): To see if BNT314 in combination with BNT327 and standard of care (SoC) chemotherapy is safe for participants and to find out the right dose of BNT314 that can be used in Part C.
* Part C (Phase 2, randomization against SoC): To see whether BNT314 and BNT327, given in combination with the usual SoC chemotherapy treatment, can shrink tumors or slow down their growth.

The study consists of a screening period, a treatment period, a safety follow-up period, and a long-term survival follow-up period.

The sponsor plans to proactively assess participant safety on a regular basis for the duration of the study according to a predefined internal review committee. In addition, an independent data monitoring committee will be developed to provide medical oversight over Part C of the study.

Participants in the study will continue to receive treatment until their disease worsens, they can no longer tolerate the treatment, or the study ends. They are expected to be on treatment for about of 6-10 months on average. After that, they will be monitored for their survival and any potential long-term side effects even after they stop participating in the study.

ELIGIBILITY:
Key Inclusion Criteria:

* Have unresectable histologically confirmed adenocarcinoma of the colon or rectum.
* Have confirmed non-microsatellite instability-high (non-MSI-H)/pMMR mCRC per Food and Drug Administration (FDA)/European Commission (EC) approved test or based on local testing.
* Have measurable disease defined by RECIST v1.1.
* Must provide a tumor tissue sample (formalin-fixed, paraffin-embedded or tissue slides) collected before C1D1 for enrollment. A newly obtained tumor sample is preferred. If it is not feasible to obtain a recent tumor sample, participants can provide archival tumor tissue (less than 2 years prior treatment).
* Have Eastern Cooperative Oncology Group Performance Status of 0 or 1.
* Have a life expectancy of ≥12 weeks.
* Have an adequate organ and bone marrow function within ≤7 days of Day 1 as defined in the protocol.
* Have had an adequate previous treatment washout period before randomization/enrollment as defined in the protocol.

Inclusion criteria applicable to only protocol-specific cohorts:

* Have received at least two previous lines of therapy for metastatic disease.
* Have progressed following first-line chemotherapy as specified in the protocol.
* Have not received prior systemic therapy for MSS/pMMR mCRC. Participants who received chemotherapy, radiotherapy, or chemoradiotherapy with curative intent for non-metastatic disease in the neoadjuvant or adjuvant setting are eligible for the study if therapy was completed at least 6 months prior to initiation of study treatment.

Other cohort-specific inclusion criteria apply.

Key Exclusion Criteria:

* Confirmed MSI-H/deficient mismatch repair mCRC (per FDA/CE approved test or based on local testing).
* Prior treatment with epithelial cell-adhesion molecule or 4-1BB targeted or immunotherapy.
* Prior treatment with immune checkpoint inhibitors or programmed death-ligand 1 (PD[L]-1)/vascular endothelial growth factor bispecific antibody.
* Is a candidate to locoregional treatment (including surgical resection, stereotactic radiation therapy or tumor ablation) with potential to induce complete or near complete response and prolonged tumor control (sometimes described as "radical" intent), per investigator's assessment.
* Have uncontrolled or significant cardiovascular disease as specified in the protocol.
* Have left ventricular ejection fraction <50% by echocardiogram within 28 days before randomization/enrollment.
* Have clinically uncontrolled pleural effusion, ascites or pericardial effusion requiring drainage, peritoneal shunt, or cell-free concentrated ascites reinfusion therapy within 2 weeks prior to randomization/enrollment.
* Have clinically active central nervous system metastases, defined as untreated and symptomatic, or requiring therapy with corticosteroids or anticonvulsants to control associated symptoms. Participants with treated brain metastases that are no longer symptomatic and who require no treatment with corticosteroids or anticonvulsants may be included in the study if they have recovered from the acute toxic effect of radiotherapy. Participants with untreated, asymptomatic brain metastasis for whom local therapy is not indicated per SoC may be eligible if neurologically stable and (if deemed necessary by the investigator). Participants at imminent risk for spinal cord compression or leptomeningeal disease are not eligible.
* Have unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet resolved to Grade ≤1 or baseline toxicities that have resolved with sequelae (e.g., tracheostomy, chronic use of feeding tube, replacement hormones) are allowed, if not associated with increased risk of complications per investigator's assessment.
* Participants in Part B or C who fulfill one of the conditions:

  * Prior treatment with anticancer therapies (as defined in the protocol) with unusual toxicity, or
  * Known dihydropyrimidine dehydrogenase (DPD) deficiency, testing performed according to the local guidelines. If not tested, lack of DPD activity must be tested for the participants who have not received anticancer therapies (as defined in the protocol) in the prior lines of treatment; testing should be performed according to the local guidelines.
* Have a history of another primary malignancy within 2 years, except adequately resected non-melanoma skin cancer, curatively treated in-situ disease, or other solid tumors curatively treated (adjuvant hormone therapy for malignancies at low risk of relapse is allowed) or have a known additional malignancy that is progressing or requires treatment.
* Have a history of small bowel obstruction requiring hospitalization within the past 3 months prior to the first dose of IMP.
* Have 24-h urine protein excretion ≥1 g. If qualitative urine protein is ≤1+, a 24-h urine protein quantitative test is not required.
* Have history of autoimmune disease (myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, psoriatic arthritis, inflammatory bowel disease, vasculitis, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, or multiple sclerosis) with a risk of exacerbation following PD-L1 inhibition or have an immune deficiency (allogeneic hematopoietic stem cell transplantation or organ transplantation). Participants with protocol-specified conditions may be eligible.
* Have serious non-healing wounds, ulcers, or bone fractures. This includes history of abdominal fistula, gastrointestinal perforation, or intra abdominal abscess or esophageal and gastric varices, acute gastrointestinal bleeding for which an interval of 6 months must pass before enrollment into this study. In addition, the participant must have undergone correction (or spontaneous healing) of the perforation/fistula and/or the underlying process causing the fistula/perforation.
* Have evidence of major coagulation disorders or other significant risks of hemorrhage.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 482 (Estimated)
Dates: Start 2025-07-18 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2031-05 (Estimated)

PRIMARY OUTCOMES:
Phase I - Part A: Occurrence of dose limiting toxicities (DLTs) during the DLT observation period | Up to 28 days after Day 1, Cycle 1
Phase I - Part A: Occurrence of treatment emergent adverse events (TEAEs) and treatment related adverse events (TRAEs) | From initiation of the first dose of BNT314 + BNT327 until 90 days after last dose of investigational medicinal product (IMP)
  Assessed according to Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0) including Grade ≥3, serious, fatal TEAEs by relationship
Phase I - Part A: Occurrence of dose interruption or discontinuation of study treatment due to TEAEs | From initiation of the first dose of BNT314 + BNT327 until 90 days after last dose of IMP
Phase I - Part B: Occurrence DLTs during the DLT observation period for the first five participants in each dose cohort | Up to 42 days after Day 1, Cycle 1
Phase I - Part B: Occurrence of TEAEs and TRAEs | From initiation of the first dose of BNT314 + BNT327 + SoC chemotherapy until 90 days after last dose of IMP
  Assessed according to CTCAE v5.0 including Grade ≥3, serious, fatal TEAEs by relationship
Phase I - Part B: Occurrence of dose interruption or discontinuation of study treatment due to TEAEs | From initiation of the first dose of BNT314 + BNT327 + SoC chemotherapy until 90 days after last dose of IMP
Phase I - Part B: Objective response rate (ORR) | From the time of initiation of the first dose of IMP to end of study, up to 57 months
  Defined as the percentage of participants in whom a complete response (CR) or confirmed partial response (PR) (assessed by the blinded independent central review [BICR] per Response Evaluation Criteria in Solid Tumors version 1.1 [RECIST v1.1]) is observed as best overall response.
Phase II - Part C: Progression free survival | From the time of initiation of the first dose of IMP to end of study, up to 57 months
  Defined as the time from randomization to first documented tumor progression (progressive disease assessed by BICR per RECIST v1.1), or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Phase II - Part C: ORR | From the time of initiation of the first dose of IMP to end of study, up to 57 months
  Defined as the percentage of participants in whom a confirmed CR or PR (assessed by BICR per RECIST v1.1) is observed as best overall response
Phase I - Part A: ORR | From the time of initiation of the first dose of IMP to end of study, up to 57 months
  Defined as the percentage of participants in whom a confirmed CR or PR (assessed by BICR per RECIST v1.1) is observed as best overall response
All parts: Duration of response | From the time of initiation of the first dose of IMP to end of study, up to 57 months
  Defined as the time from first objective response (CR or PR assessed by BICR per RECIST v1.1) to first occurrence of objective tumor progression (progressive disease assessed by BICR per RECIST v1.1) or death from any cause, whichever occurs first.
Phase I - Part A and Part B: Disease control rate | From the time of initiation of the first dose of IMP to end of study, up to 57 months
  Defined as the percentage of participants with confirmed CR or PR or stable disease (per RECIST v1.1, assessed at least 6 weeks after the first IMP dose) observed as best ORR per BICR.
Phase I - Part A and Part B: Geometric mean of pharmacokinetic parameter maximum concentration of BNT314 and BNT327 in serum | From predose to 42 days after first dose of IMP
  Per dose level. If data permits.
Phase I - Part A and Part B: Geometric mean of pharmacokinetic parameter time taken to reach maximum concentration of BNT314 and BNT327 in serum | From predose to 42 days after first dose of IMP
  Per dose level. If data permits.
Phase I - Part A and Part B: Geometric mean of pharmacokinetic parameter half life of BNT314 and BNT327 in serum | From predose to 42 days after first dose of IMP
  Per dose level. If data permits.
Phase I - Part A: Geometric mean of pharmacokinetic parameter volume of distribution of BNT314 and BNT327 in serum | From predose to 42 days after first dose of IMP
  Per dose level. If data permits.
Phase I - Part A: Geometric mean of pharmacokinetic parameter area under the curve of BNT314 and BNT327 in serum | From predose to 42 days after first dose of IMP
  Per dose level. If data permits.
Phase I - Part A and Part B: Geometric mean of pharmacokinetic parameter clearance of BNT314 and BNT327 in serum | From predose to 42 days after first dose of IMP
  Per dose level. If data permits.
Phase I - Part B: Geometric mean of pharmacokinetic parameter steady state volume of distribution of BNT314 and BNT327 in serum | From predose to 42 days after first dose of IMP
  Per dose level. If data permits.
Phase I - Part B: Geometric mean of pharmacokinetic parameter total drug exposure across time of BNT314 and BNT327 in serum | From predose to 42 days after first dose of IMP
  Per dose level. If data permits.
Phase I - Part B: Geometric mean of pharmacokinetic parameter area under the concentration-time curve from pre-dose to last quantifiable time point prior to the next dose of BNT314 and BNT327 in serum | From predose to 42 days after first dose of IMP
  Per dose level. If data permits.
Phase I - Part A and Part B: ADA prevalence | Up to 90 days post last dose of IMP
  Percentage of participants who are ADA positive (either baseline or post-baseline). By dose level. If data permits.
Phase I - Part A and Part B: Anti-drug antibody (ADA) incidence | Up to 90 days post last dose of IMP
  Percentage of participants having treatment-emergent ADA. By dose level. If data permits.
Phase II - Part C: Overall survival | From the time of initiation of the first dose of IMP to end of study, up to 57 months
  Defined as the time from randomization to death from any cause
Phase II - Part C: Occurrence of TEAEs and TRAEs | From initiation of the first dose of BNT314 + BNT327 until 90 days after last dose of IMP
  Assessed according to CTCAE v5.0 including Grade ≥3, serious, fatal TEAEs by relationship
Phase II - Part C: Occurrence of dose interruption or discontinuation of study treatment due to TEAEs | From initiation of the first dose of BNT314 + BNT327 until 90 days after last dose of IMP

CONTACTS AND LOCATIONS:
Overall Officials: BioNTech Responsible Person, Study Director — BioNTech SE
Locations (7):
- United States (3):
  - START Midwest, Grand Rapids, Michigan
  - Cleveland Clinic Taussig Cancer Institute Case Comprehensive Cancer Center, Cleveland, Ohio
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Spain (2):
  - Hospital HM Nou Delfos, Barcelona
  - Centro Integral Oncologico Clara Campal, Madrid
- United Kingdom (2):
  - Guy's & St Thomas' NHS Foundation Trust, Guy's Hospital, London
  - The Royal Marsden NHS, Sutton

IPD SHARING:
Plan to Share IPD: No